CLINICAL TRIAL: NCT04835064
Title: A Phase III, Multicenter, Prospective, Randomized, Patients With Resectable Pancreatic Cancer With Elevated Serum CA125 Were Compared With Those Who Did Not Receive Neoadjuvant Chemotherapy.
Brief Title: Pancreatic Cancer With Elevated Serum CA125 Were Compared With Those Who Did Not Receive Neoadjuvant Chemotherapy.
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Fudan University (Other)
Responsible Party: Principal Investigator, Xian-Jun Yu, President of Shanghai Pancreatic Cancer Institute, Fudan University
Allocation: Non-Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: CSPAC-4
Record Dates: First submitted 2021-04-02; First posted 2021-04-08 (Actual); Last update posted 2021-04-08 (Actual); Status verified 2021-04

CONDITIONS: Pancreatic Adenocarcinoma
MeSH Terms: interventions — Taxes; Albumin-Bound Paclitaxel; Gemcitabine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Nab-paclitaxel and Gemcitabine (Experimental): Albumin combined with paclitaxel 125mg/m2 intravenous infusion, Day 1, 8, 15;Gemcitabine 1000 mg/m2 was given intravenously for more than 30min on days 1, 8, and 15, and repeated every 4 weeks.
  Interventions: Drug: Nab paclitaxel; Drug: Gemcitabine
- mFOLFIRINOX (Experimental): Oxaliplatin 85 mg/m2 intravenous infusion for 2 h, Day 1;LV 400 mg/m2 intravenous infusion for 2 h, Day 1;Irinotecan 150 mg/m2 was added 30 min after intravenous infusion for 90 min, day 1;This was immediately followed by a continuous intravenous infusion of 5-FU 2400 mg/m2 for 46 h.Repeat every 2 weeks.
  Interventions: Drug: mFOLFIRINOX

INTERVENTIONS:
Drug: Nab paclitaxel — Albumin combined with paclitaxel 125mg/m2 intravenous infusion, Day 1, 8, 15
  Other Names: Abraxane
  Arms: Nab-paclitaxel and Gemcitabine
Drug: Gemcitabine — Intravenous infusion of 1000 mg/m2 was given for more than 30min on days 1, 8, and 15, and repeated every 4 weeks
  Other Names: Gemzar
  Arms: Nab-paclitaxel and Gemcitabine
Drug: mFOLFIRINOX — Oxaliplatin 85 mg/m2 intravenous infusion for 2 h, Day 1;LV 400 mg/m2 intravenous infusion for 2 h, Day 1;Irinotecan 150 mg/m2 was added 30 min after intravenous infusion for 90 min, day 1;This was immediately followed by a continuous intravenous infusion of 5-FU 2400 mg/m2 for 46 h.Repeat every 2 weeks.
  Other Names: modified FOLFIRINOX regimen
  Arms: mFOLFIRINOX

SUMMARY:
The main purpose of

* To observe the overall survival of patients with resectable pancreatic cancer with elevated serum CA125 with and without neoadjuvant chemotherapy A secondary purpose
* To observe relapse-free survival in patients with resectable pancreatic cancer with elevated serum CA125 versus without neoadjuvant chemotherapy
* To observe the resectable rate of patients with resectable pancreatic cancer with elevated serum CA125 with and without neoadjuvant chemotherapy
* To observe the safety parameters of patients with resectable pancreatic cancer with or without neoadjuvant chemotherapy with elevated serum CA125

DETAILED DESCRIPTION:
This study is a prospective, multicenter, randomized, controlled Ⅲ period clinical trials.A total of 600 patients with resectable pancreatic cancer assessed by imaging and serum CA125≥35 U/mL were randomly assigned according to the ratio of 1:1 (300 cases: 300 cases) between the direct surgical resection group and the neoadjuvant chemotherapy group, to observe the efficacy and safety of patients with resectable pancreatic cancer with elevated serum CA125 with or without neoadjuvant chemotherapy.Neoadjuvant chemotherapy and adjuvant chemotherapy can use albumin-binding paclitaxel combined with gemcitabine (AG) regimen or mFOLFirinox (5-FU, calcium leucofolate [LV], irinotecan, oxaliplatin) regimen. AG regimen was given on day 1, 8, 15, and repeated every 4 weeks.The mFOLFIRINOX regimen was administered on days 1 and 15 and repeated every 4 weeks.Patients in the neoadjuvant chemotherapy group were treated with 4 courses of neoadjuvant chemotherapy (AG regimen or mFOLFIRINOX regimen) immediately after the pathologic diagnosis of pancreatic adenocarcinoma was confirmed by puncture.Patients receiving neoadjuvant chemotherapy will undergo surgical exploration to assess the resectability of the tumor.Four to eight weeks after radical resection, the patients were treated with adjuvant chemotherapy from the recovery of surgical trauma. The choice of adjuvant chemotherapy after surgery depended on the response to neoadjuvant chemotherapy.If neoadjuvant chemotherapy is effective, adjuvant chemotherapy will maintain the original regimen;If neoadjuvant chemotherapy is ineffective but radical surgery is still feasible, adjuvant chemotherapy will be used with a crossover regimen.Neoadjuvant chemotherapy group received adjuvant chemotherapy for 2 courses.In the direct surgical resection group, 6 courses of adjuvant chemotherapy were started 4 to 8 weeks after radical resection.Relevant examinations should be conducted before and after each course of medication to evaluate safety events. Imaging reexaminations should be conducted every 2 courses of medication, and imaging reexaminations should be conducted every 3 months during follow-up to evaluate disease recurrence.

ELIGIBILITY:
Inclusion Criteria:

1. Voluntarily participate and sign the informed consent;
2. Age ≥18 years old and ≤75 years old, no gender limitation;
3. ECOG score ≤1;
4. Imaging evaluation of resectable pancreatic cancer, serum CA125≥35 U/mL;
5. pancreatic adenocarcinoma confirmed by pathology after pancreatic puncture or surgery;
6. No distant metastasis, malignant abdominal effusion or pleural effusion before neoadjuvant chemotherapy;Postoperative baseline chest, abdomen and pelvis CT showed no tumor metastasis/recurrence.
7. Expected survival ≥3 months;
8. No serious hematopoietic dysfunction, abnormal functions of heart, lung, liver and kidney and immune deficiency were observed. The laboratory test results met the following criteria: blood routine indicators: white blood cell (WBC) ≥3×109/L;Absolute neutrophils count (ANC) ≥1.5×109/L;Platelet (PLT) ≥100×109/L;Hemoglobin (HGB) ≥9g/dL;Blood biochemical indexes: AST (SGOT), ALT (SGPT) ≤2.5× upper limit of normal value (ULN);Total bilirubin (TBil) ≤ULN;Serum creatinine (CRE) ≤1.5×ULN;Coagulation function: Prothrombin time (PT), international standardized ratio (INR) ≤1.5×ULN;
9. the willingness of women with potential fertility to use medically approved contraceptives in the trial;
10. Able to follow the research visit plan and other program requirements.

Exclusion Criteria:

1. Patients had received any type of anti-tumor therapy before enrolment, including interventional chemoembolization, ablation, radiotherapy, chemotherapy, and molecular targeted therapy;
2. have central nervous system diseases, mental diseases, unstable angina pectoris, congestive heart failure, severe arrhythmia and other uncontrollable serious diseases;
3. Uncontrolled infection, bleeding, pancreatic leakage, bile leakage, or other postoperative complications at baseline;Acute and chronic metabolic acidosis (including ketoacidosis and lactic acidosis) cannot be corrected;
4. Have a history of other malignant tumor diseases;
5. Have a history of allergy to the study drug or similar drug structure;
6. Pregnant and lactating women;
7. Other reasons why the investigator considers it inappropriate to participate in the clinical study.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 600 (Estimated)
Dates: Start 2021-04-01 (Estimated); Primary Completion 2024-04-01 (Estimated); Study Completion 2024-12-01 (Estimated)

PRIMARY OUTCOMES:
overall survival | from randomization to death, up to 36 months
  • To observe the overall survival of patients with resectable pancreatic cancer with elevated serum CA125 with and without neoadjuvant chemotherapy

SECONDARY OUTCOMES:
Relapse-free survival | from randomization to recurrence, up to 36 months
  To observe the relapse-free survival of patients with resectable pancreatic cancer with elevated serum CA125 versus without neoadjuvant chemotherapy
Surgical excision rate | from randomization to recurrence, up to 36 months
  • To observe the resectable rate of patients with resectable pancreatic cancer with elevated serum CA125 with and without neoadjuvant chemotherapy
Incidence of adverse events | from randomization to recurrence, up to 36 months
  • To observe the Incidence of adverse events of patients with resectable pancreatic cancer with or without neoadjuvant chemotherapy with elevated serum CA125

CONTACTS AND LOCATIONS:
Overall Officials: Xian-Jun Jun, M.D., Ph.D., Principal Investigator — Fudan University

IPD SHARING:
Plan to Share IPD: No